CLINICAL TRIAL: NCT04395339
Title: Ganglioside-Monosialic Acid Prophylaxis for Cognitive Dysfunction Related to Whole Brain Radiotherapy in Breast Cancer Patients With Brain Metastases ，a Multi-center，Randomized，Single Blind，Phase III Clinical Trail
Brief Title: GM1 Prophylaxis for WBRT Related Cognitive Dysfunction
Acronym: GLORY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSUCC-012
Record Dates: First submitted 2020-05-06; First posted 2020-05-20 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Brain Metastases; Radiotherapy Side Effect; Cognitive Impairment; Gangliosidosis, GM1; Breast Cancer
Keywords: WBRT; Gangliosidoses; Brain Metastases; radiotherapy; breast cancer
MeSH Terms: conditions — Brain Neoplasms; Radiation Injuries; Cognitive Dysfunction; Gangliosidosis, GM1; Breast Neoplasms; Gangliosidoses | interventions — G(M1) Ganglioside; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm(GM1) (Experimental): This arm will be treated with GM1.
  Interventions: Drug: Monosialotetrahexosyl ganglioside (GM1)
- Control arm (Placebo Comparator): This arm will be treat with blank placebo.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Monosialotetrahexosyl ganglioside (GM1) — Ganglioside-Monosialic Acid is added into 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 15 days. The first dose is given at 1 day before the start of the radiotherapy.
  Other Names: a group of galactose-containing cerebrosides found in the surface membranes of nerve cells
  Arms: Experimental arm(GM1)
Drug: Control — 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 15 days. The first dose is given at 1 day before the start of the radiotherapy.
  Other Names: 0.9% sodium chloride
  Arms: Control arm

SUMMARY:
To evaluate the efficacy and safety of GM1 for preventing cognitive impairment related to whole brain radiotherapy in breast cancer patients with brain metastases. And explore the clinical and molecular parameter for predicting severe cognitive impairment induced by WBRT and gaining benefit from GM1.

Primary Endpoint: the change of Hopkins Verbal and Learning Test-Revised Delayed Recall,HVLT-R DR,before and after WBRT Secondary ENDPOINT: the change of Alzheimer's Disease Assessment Scale-Cognitive，ADAS-Cog before and after WBRT;severe cognitive impairment percentage and onset time; Design:204 patients will be randomly assigned to exp.group,102 cases,and 102 cases of control group.

DETAILED DESCRIPTION:
Background:Brain metastasis is a common event for advanced stage cancer,and whole brain radiotherapy(WBRT)is one of the most effective and widely utilized measures for brain metastases.Gaining control of the brain metastases may provide better survival for patients,but can also cause cognitive impairment,sometimes may be severe.Considering cognitive function is one of the most important aspect of quality of life(QoL), some remedies for the treatment-related adverse effect should be provided. Some agents were evaluated for this purpose,and results were unsatisfying. Ganglioside-Monosialic Acid (GM1) is used as an neuroprotective agent after brain surgery or neurodegenerative disease,and a clinical trail(NCT02468739) hosted by our team demonstrated that it could relief taxane-induced neurotoxicity.So GM1 is proposedto be effective in treating WBRT related cognitive dysfunction.

Outline:This will be an single-blind,randomized study,102 patients planning to receive WBRT will be allocated to control and experiment group,respectively,to receive GM1(100mg D0-D14) or placebo(0.9% saline).Cognitive scales will be utilized to evaluate the efficacy.

PRIMARY OBJECTIVE:

Evaluate the efficacy of GM1 in alleviating WBRT related cognitive impairment by Hopkins Verbal and Learning Test Revised-Delayed Recall(HVLT-R DR) before and after RT.

Secondary Objective:

Evaluate the efficacy of GM1 in alleviating WBRT related cognitive impairment by Alzheimer's Disease Assessment Scale-Cognitive(ADAS-Cog )before and after RT.

Evaluate the efficacy of GM1 in alleviating WBRT related cognitive impairment by Mini-mental state Examination(MMSE)before and after RT.

Evaluate the efficacy of GM1 in alleviating WBRT related cognitive impairment by comparing severe cognitive impairment incidence,and onset time of cognitive dysfunction.

Explore the molecular parameter for GM1 benefit. Treatment group: Ganglioside-Monosialic Acid is added into 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 15 days. The first dose is given at 1 day before the start of the radiotherapy. At the same time, the patients are treated with a WBRT protocol selected by the investigators.

Placebo group: Placebo is 250 mL of 0.9% sodium chloride injection, which is given once a day via intravenous drip infusion for 15 days. The first dose is given at 1 day before the start of the RT. At the same time, the patients are treated with a WBRT protocol selected by the investigators.

Follow up: Assessment will be performed before and 12,24 36,48 weeks after RT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75,with histological affirmative breast cancer ,and over 4 brain metastases ,need for WBRT suggested by radiotherapy oncologist ;
* Estimated survival time over 6months;
* Abundant hematological function:Absolute Neutrophil Count≥2×109/L ;platelet count≥100×109/L and hemoglobulin≥9 g/dL;
* Abundant liver function：total bilrubin≤ULN；ASTandALT≤2.5ULN；AKP≤5ULN
* Can cope with HVLT-RDR and ADAS-Cog evaluation
* No prior therapy could induce neurological damage,within 4 weeks
* No more that 1 degree peripheral neuropathy or any other diseases or symptoms that could hinder the evaluation of neurological AE
* No more treatment or nursing is allowed after enrolling this trail
* Written Informed Consent signed

Exclusion Criteria:

* PS score over 2,and estimated no attenuation by WBRT
* Women with pregnancy or breast feeding
* Unwilling to contraception measurement
* Abnormal baseline impairment of cognitive impairment
* Allergy to experiment agents or components
* Unsuitable to GM1 treatment, evaluated by investigators
* Active infection
* RT dose over 30Gy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
HVLT R-DR | 24 weeks after WBRT.
  The change of score for Hopkins verbal learning test -revised,delayed recall,form baseline to 24weeks after WBRT,score ranges from 0 to 12,higher score indicates better cognitive function

SECONDARY OUTCOMES:
ADAS-Cog | 24 weeks after WBRT.
  The change of score for Alzheimer's Disease Assessment Scale-Cognitive，ADAS-Cog,form baseline to 24 weeks after WBRT,score ranges from 0 to 75,LOWER score indicates better cognitive function
MMSE | 24 weeks after RT.
  The change of score for Minimal Mental State Examination,MMSE,form baseline to 24 weeks after WBRT,higher score indicates better cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No